CLINICAL TRIAL: NCT02159313
Title: Relative Bioavailability Study of Riociguat Given Orally as a Crushed 2.5 mg Tablet Suspended in Applesauce, Crushed 2.5 mg Tablet Suspended in Water, and Whole 2.5 mg Tablet After a Continental Breakfast in Comparison to a Whole 2.5 mg Tablet Given in the Fasted State to Characterize the Pharmacokinetic Properties in Healthy Male Adult Subjects in a 4-fold Crossover Design
Brief Title: Relative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 17306; 2013-005166-18 (EudraCT Number)
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Healthy Volunteers
Keywords: Biological Availability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BAY63-2521 with Non sparkling water (Experimental): Single dose of a whole 2.5 mg riociguat tablet (fasted) with 240 mL of non-sparkling water at room temperature
  Interventions: Drug: Riociguat(Adempas,BAY63-2521)
- BAY63-2521 with applesauce (Experimental): Single dose of a crushed 2.5 mg riociguat tablet suspended in 50 mL applesauce, to be eaten with a spoon (fasted)
  Interventions: Drug: Riociguat(Adempas,BAY63-2521)
- BAY63-2521 with water (Experimental): Single dose of a crushed 2.5 mg riociguat tablet suspended in a glass with 25 mL water, to be drunk and flushed twice with 25 mL water in the same glass (fasted)
  Interventions: Drug: Riociguat(Adempas,BAY63-2521)
- BAY63-2521 after breakfast (Experimental): Single dose of a whole 2.5 mg riociguat tablet taken within 5 minutes after the last bite of a continental breakfast (fed) with 240 mL of non-sparkling water at room temperature
  Interventions: Drug: Riociguat(Adempas,BAY63-2521)

INTERVENTIONS:
Drug: Riociguat(Adempas,BAY63-2521) — Single dose of a whole 2.5 mg riociguat tablet

SUMMARY:
To investigate relative bioavailability of crushed tablets suspended in apple sauce or water

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 45 years (inclusive) at the first screening examination
* Ethnicity: white
* Body mass index (BMI): >18 and <29.9 kg/m2

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, or effects of the study drug will not be normal
* History of coronary artery disease
* Symptomatic postural hypotension (e.g. dizziness, lightheadedness)
* History of bronchial asthma or any other airway disease
* Smoking (former smokers who have stopped smoking at least 3 months before the first study drug administration may be included)
* Clinically relevant findings in the ECG such as a second- or third-degree atrioventricular block, prolongation of the QRS complex over 120 ms or of the QTc interval (QT interval corrected for heart rate) over 450 ms
* Systolic blood pressure below 100 or above 145 mmHg
* Diastolic blood pressure below 50 or above 95 mmHg
* Heart rate below 45 or above 95 beats per minute

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of riociguat in plasma by Area under the plasma concentration time curve (AUC) | Multiple time points up to day 3
Pharmacokinetics of riociguat in plasma by maximal concentration (Cmax) | Multiple time ponits up to day 3

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mönchengladbach, North Rhine-Westphalia, Germany